CLINICAL TRIAL: NCT04015726
Title: Secular Trends in the Prevalence of Cardiometabolic Risk Factors Among Teenage School Children in Urban South India
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: IDRFARH012
Record Dates: First submitted 2019-06-29; First posted 2019-07-11 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Dysglycemia; Dyslipidemias; Hypertension; Insulin Resistance
MeSH Terms: conditions — Obesity; Dyslipidemias; Hypertension; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of cardiometabolic risk is high among South Asians which manifests itself at an early age. Studies have reported that unhealthy food choices, inadequate physical activity and lack of awareness on healthy lifestyle practices pose a huge threat to the increasing prevalence of metabolic abnormalities even at adolescence. In an earlier study conducted in 2006, reported that 68% of the children during their early adolescence had one or more of the cardiometabolic abnormalities such as obesity, central adiposity, increased blood pressure and presence of dysglycaemia and dyslipidaemia. The risk escalated with increasing weight. Therefore, it is imperative to sensitize the children on improving their lifestyle by conducting screening tests and health education programmes in schools by involving teachers. The Investigator have also shown in a study that teachers can be instrumental in imparting knowledge on the prevention of non-communicable diseases such as diabetes by promoting healthy behavioral changes. The proposed study will focus on a) changes in the prevalence of cardiometabolic risk factors over a 10 year period b) health education programme to school children c) recommendations to school teachers (tool-kit) to inculcate improved lifestyle practices to their students.

DETAILED DESCRIPTION:
This programme will be conducted after obtaining prior permission from the Directorate of School Education, Government of Tamil Nadu and school authorities. This study will be conducted in 22 schools in Chennai involving 2815 students of age group 12 to 18 years. Initially the study and its procedure will be explained to the principal and the teachers of the school. Request the school authority to fix a date for each standard/grade to explain about the informed consent / assent form and the study process to the students. The students will be asked to give the informed consent/assent form to their parents and asked to get their signature in the specified place. Instruction will be given to the students that their parents can call the Investigator if they have any doubts in the informed consent/assent form. After giving ample time for the informed consent process the students will be asked to give the informed consent when the research team goes to the school. The informed consent should be countersigned by the teachers to confirm the authenticity of the parent's signature. The research team gets the signature from the student in the assent form. A date is finalized with the school authority for the screening. The students are advised to come in fasting for the test. On the day of screening the student will be given a screening number. Necessary details such as personal and family information, anthropometry (height, weight, waist circumference, body fat) and blood pressure will be measured. Medical history, diet, physical activity, and sleep habits and questionnaire on awareness on diabetes will be recorded. Laboratory investigations such as fasting blood glucose, plasma insulin and lipid profile (Total Cholesterol, Triglyceride, Low-Density Lipoprotein (LDL), Very Low-Density Lipoprotein (VLDL) and High-Density Lipoprotein (HDL)) will be measured.

After the assessment, the students will be given refreshments and a few minutes of rest. The samples will be sent to the central laboratory for analyses. The reports will be distributed to the students within a week's time. Parents will be personally contacted by the research team if there is any concern in the lab report which requires medical attention.

ELIGIBILITY:
Inclusion Criteria:

1. Children both boys and girls between 12 - 18yrs age group
2. Parents and child willing to give informed consent
3. Children must be available for and willing to attend all evaluation visits
4. Willingness to follow the protocol requirements as evidenced by written informed consent

Exclusion Criteria:

1. Children below the age of 12 years and above the age of 18 years
2. Parents or Child who is not willing to participate in the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children both boys and girls between 12 - 18yrs age group
Sampling Method: Non-Probability Sample
Enrollment: 2815 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of central adiposity | baseline
  Among adolescent children in 2019 in comparison with 2006 data
Prevalence of dysglycemia | Baseline
  Among adolescent children in 2019 in comparison with 2006 data
Prevalence of dyslipidemia | Baseline
  Among adolescent children in 2019 in comparison with 2006 data
Prevalence of hypertension | Baseline
  Among adolescent children in 2019 in comparison with 2006 data
Prevalence of insulin resistance | Baseline
  Among adolescent children in 2019 in comparison with 2006 data

SECONDARY OUTCOMES:
Prevalence of overweight | Baseline
  Among adolescent children in 2019 in comparison with 2006 data
Prevalence of obesity | Baseline
  Among adolescent children in 2019 in comparison with 2006 data
Changes in diet habit | Baseline
  Among adolescent children in 2019 in comparison with 2006 data
Changes in duration of physical activity | Baseline
  Among adolescent children in 2019 in comparison with 2006 data

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, MD, PhD, DSc, Principal Investigator — Senior Research Officer
Locations (1):
- India Diabetes Research Foundation, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Undecided